CLINICAL TRIAL: NCT06698835
Title: The Effect of Turnip Consumption and Qigong Exercise Program on Weight Loss Among Female Students: Clinical Trail
Brief Title: Turnip Consumption and Qigong Exercise Program on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: King Faisal University (Other)
Responsible Party: Principal Investigator, Safaa Rabea Osman, assistant professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: turnip& qigong exercise
Record Dates: First submitted 2024-02-09; First posted 2024-11-21 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Obesity, Adolescent
Keywords: obesity; qigong exercise; turnip consumption; weight loss
MeSH Terms: conditions — Pediatric Obesity; Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: the study design indicates two arms (e.g., experimental and control) which will divide the group into small groups (5 in each) for experimental. and 10 students as a control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- school girls aged 10-12 years (case group) (Experimental): It includes turnip consumption, and qigong exercise. Also, they will receive health education about the importance of weight loss. Educational program aged from 10 to 12 years. they will receive the nursing educational program which will be implemented in 2 small groups (5) in the primary school
  Interventions: Dietary Supplement: Turnip Consumption
- school girls aged 10-12 years (control group) (No Intervention): it includes ten students as control group who will not receive any intervention

INTERVENTIONS:
Dietary Supplement: Turnip Consumption — Turnip Consumption and Qigong Exercise with educational Program about loss of weight
  Other Names: Qigong Exercise
  Arms: school girls aged 10-12 years (case group)

SUMMARY:
Obesity and weight-related issues are prevalent concerns affecting individuals worldwide, with particular significance among the younger demographic, such as female students. As lifestyles evolve and dietary habits play a pivotal role in overall well-being, exploring innovative approaches to weight management becomes imperative. Thus, obesity is a huge public health importance with economic emotional and social consequences.

DETAILED DESCRIPTION:
Obesity is an epidemic causing serious health consequences, including diabetes, dyslipidemia, and hypertension. Obesity in adolescents can cause chronic brain hypoxia and affect learning. Weight loss occurs when energy intake is less than energy expenditure, and achieving an energy deficit remains the main dietary target. The evidence for the specific impact of vegetables is qualified. Recently, there has been much scientific interest and debate on the potential link between dairy consumption and body weight regulation. The idea of turnip consumption and qigong exercise includes a broad variety of subjects. vegetables are high in water and fiber and low in energy density, so their consumption is suggested to prevent obesity. Moreover, Traditional Chinese exercises are an ancient way of exercise and fitness, which have been reported to have unique advantages in the treatment of obesity.

ELIGIBILITY:
Inclusion Criteria:

* aged from 10 to 12 years
* free from any chronic diseases
* accept to participate

Exclusion Criteria:

* have any digestive problems
* unable to communicate or participate

Ages: 10 Years to 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
change fat mass index | 3 months
  it will be measured before and after the program
weight loss | 3 months
  It will be assessed by Body mass index before and after applying the intervention (Turnip Consumption and Qigong Exercise) and measure their effect on weight

SECONDARY OUTCOMES:
assess their endurance | 3 months
  by using Harvard Step Test before and after the intervention (is a test of aerobic fitness, developed by Brouha et al. (1943) in the Harvard Fatigue Laboratories during WWII)
pulse Rate | 2 weeks
  by assessing pulse before and after the intervention
respiration rate | 2 weeks
  measure respiration rate before and after intervention
heart rate | 2 weeks
  measure heart rate before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Safaa Osman, Principal Investigator — Egypt- faculty of nursing
Locations (1):
- Faculty of Nursing, Asyut, Egypt